CLINICAL TRIAL: NCT01981590
Title: Mapping for Acute Transvenous Phrenic Nerve Stimulation Study (MAPS Study)
Brief Title: Mapping for Acute Transvenous Phrenic Nerve Stimulation Study
Acronym: MAPs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic BRC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAPs-breathing
Record Dates: First submitted 2013-09-20; First posted 2013-11-11 (Estimated); Results first posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-02

CONDITIONS: Sleep Apnea
Keywords: breathing, heart failure, sleep apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Respiratory Aspiration; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All enrolled patients (Experimental): All enrolled patients that underwent a scheduled cardiac catheterization involving an atrial fibrillation (AF) ablation procedure as per clinical practice
  Interventions: Device: Stimulating the phrenic nerve intravenously using high frequency electrical pulses using an EP catheter connected to external pulse stimulator.

INTERVENTIONS:
Device: Stimulating the phrenic nerve intravenously using high frequency electrical pulses using an EP catheter connected to external pulse stimulator. — Intravenously stimulating the phrenic nerve with an EP catheter using high frequency electrical pulses as generated by the model 19039 external neurostimulator.

SUMMARY:
The Mapping for Transvenous Phrenic Nerve Stimulation Study (MAPS) is being conducted to evaluate the feasibility of transvascular stimulation of phrenic nerves via an electrophysiology (EP) catheter advanced into the great veins.

DETAILED DESCRIPTION:
Purpose The Mapping for Transvenous Phrenic Nerve Stimulation Study (MAPS) is being conducted to evaluate the feasibility of transvascular stimulation of phrenic nerves via an EP catheter advanced into the great veins.

Study Design This is a prospective, non-randomized, acute feasibility study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects older than 18 years of age
* Subject is undergoing a cardiac catheterization involving right heart catheterization and/or EP procedures and/or device implant.
* Subjects willing and able to give informed consent

Exclusion Criteria:

* Subject with a previously implanted transvenous lead, which is still present in the veins under study.
* Subject with evidence of phrenic nerve palsy.
* Subject with chronic obstructive pulmonary disease.
* Subject with a spinal cord stimulator.
* Subject needs to receive drugs that might interfere with patient perception.
* Subjects with medical conditions that would prevent study participation
* Subjects who are pregnant, nursing, or of child bearing potential and are not on a reliable form of birth control
* Subjects enrolled in concurrent studies which could confound the results of this study
* Subject is unable or unwilling to participate with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frieder Braunschweig, MD, PhD, Principal Investigator — Karolinska Institute, department of Cardiology
Locations (2):
- Stichting Catharina Ziekenhuis, Eindhoven, EJ, Netherlands
- Karolinska University Hospital, Solna, Stockholm, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 15 subjects have been enrolled, in Sweden (Karolinska University Hospital, Solna in Stockholm) and in The Netherlands (Catherina Hospital in Eindhoven).
  All the 15 subjects enrolled underwent the study procedure and performed the 2-4 weeks post-procedure assessment follow-up
Groups:
- Phrenic Nerve Stimulation: Intravenously stimulating the phrenic nerve
  Stimulating the phrenic nerve intravenously using high frequency electrical pulses using an EP catheter connected to external pulse stimulator.: Intravenously stimulating the phrenic nerve with an EP catheter using high frequency electrical pulses as generated by the model 19039 external neurostimulator.
Period: Overall Study
Arm/Group | Phrenic Nerve Stimulation
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Phrenic Nerve Stimulation
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Region of Enrollment [Number; unit: participants]
  Sweden | 7
  Netherlands | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Response to Stimulation (Diaphragmatic Movement Achieved)
Description: Number of Patients With Response to Stimulation, defined by Presence of Movement of the Diaphragm Induced by a Pacing Stimulus With Pulse Amplitude of 10 V or Less
Time Frame: one hour
Population: All 15 enrolled patients who were undergoing an atrial flutter or atrial fibrillation ablation procedure
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Phrenic Nerve Stimulation Achieved: Intravenously stimulating the phrenic nerve with an EP catheter using high frequency electrical pulses as generated by the model 19039 external neurostimulator.
Arm/Group | Patients With Phrenic Nerve Stimulation Achieved
Number analyzed (Participants) | 15
Participants | 15

2. Secondary Outcome: Number of Patients With Response to Stimulation (Tidal Volume)
Description: Number of Patients With Response to Stimulation, defined by measured tidal volume of 200 ml or more induced by a pacing stimulus with pulse amplitude of 4 V or less
Time Frame: one hour
Population: All 15 enrolled patients who were undergoing an atrial flutter or atrial fibrillation ablation procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Phrenic Nerve Stimulation Achieved
Number analyzed (Participants) | 15
Participants | 9

3. Secondary Outcome: Number of Patients With Observed Side Effects
Description: Number of patients with observed side effects like potential physiologic changes or side effects associated with transvenous nerve stimulation
Time Frame: From procedure to 2-4 weeks post-procedure
Population: All 15 enrolled patients who were undergoing an atrial flutter or atrial fibrillation ablation procedure
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Observed Side Effects: All Patients enrolled in the study that underwent an atrial flutter or atrial fibrillation ablation procedure with observed side effects
Arm/Group | Patients With Observed Side Effects
Number analyzed (Participants) | 15
Participants | 6

4. Secondary Outcome: Number of Observed Side Effects
Description: All observed side effects like potential physiologic changes or side effects associated with transvenous nerve stimulation such as pain, hiccup, skeletal muscular tremor, nausea, and sinus node activation
Time Frame: From procedure to 2-4 weeks post-procedure
Population: All 15 enrolled patients who were undergoing an atrial flutter or atrial fibrillation ablation procedure
Measure: Number; unit: Side Effect
Arm/Group | Patients With Observed Side Effects
Number analyzed (Participants) | 15
Side Effect | 7

ADVERSE EVENTS:
Time Frame: From procedure to 2-4 weeks post-procedure
Arm/Group | Phrenic Nerve Stimulation
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 4/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phrenic Nerve Stimulation (N=15)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phrenic Nerve Stimulation (N=15)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No